CLINICAL TRIAL: NCT04391712
Title: Multiwave Locked System (MLS) Laser Therapy for COVID-19 Positive Patients With Pulmonary Disease
Brief Title: Photobiomodulation Laser Therapy for COVID-19 Positive Patients With Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lowell General Hospital (Other)
Responsible Party: Principal Investigator, Scott Sigman, MD, Principal Investigator, Lowell General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.01
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID; Laser; Pulmonary
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental (Experimental): Participants will receive MLS laser treatment along with regular inpatient medical care.
  Interventions: Device: MLS Laser
- Control Group (Active Comparator): Participants will receive regular inpatient medical care.
  Interventions: Other: Regular Inpatient Medical Care

INTERVENTIONS:
Device: MLS Laser — Treatments will be delivered to the participants days 1-4, in a prone position using a 10 by 25 cm laser field across each lung with 7j/cm2 at 1500 Hz.
  Arms: Experimental
Other: Regular Inpatient Medical Care — Regular inpatient medical care
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of MLS laser therapy as a treatment for pulmonary complications due to COVID-19 infection.

DETAILED DESCRIPTION:
Participants will be randomized into treatment vs. control group. Both groups will receive regular inpatient medical treatment. Participants in the experimental arm will receive laser treatments once daily for 4 days. Treatments will be delivered to the patients in a prone position using a 10 by 25 cm laser field across each lung with 7j/cm2 at 1500 Hz. Standard nursing protocols would be used to identify participant's pulmonary status throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive
* Pulmonary compromise requiring oxygen support of approximately 2-6 liters
* Able to self prone, or support in self-sitting position

Exclusion Criteria:

* Ventilator management
* Patients with autoimmune disorders or inflammatory conditions not related to COVID-19
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Patient Disposition Post treatment | 7 days
  ICU on vent, ICU not requiring ventilation, Discharge to Rehab requiring assistance, Discharge to Home unable to perform ADL's, Discharge to Home able to perform ADL's
oxygenation | Daily for 4 days
  Patients oxygen requirements pulse oximetry will be evaluated for change from pre and post individual treatment as well as end of protocol
IL-6 levels | First four days of trial
  The change in pre treatment levels and 24 hours post final treatment
Chest Xray radiographic results | 7 Days
  Pre treatment CXR will be compared to post treatment CXR using the RALE CXR evaluation scale
Brescia-COVID Respiratory Severity Scale | 7 days
  The change in pretreatment and post treatment BCRSS will be evaluated
SMART-COP Score | 7 days
  The change in pretreatment and post treatment scores will be evaluated
PSI Score | 7 days
  The change in pretreatment and post treatment scores will be evaluated
CRP levels | 7 days
  The change in pretreatment and post treatment levels will be evaluated The change in pretreatment and post treatment levels will be evalutated

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sigman, MD, Principal Investigator — Lowell General Hospital
Locations (1):
- Lowell General Hospital, Lowell, Massachusetts, United States